CLINICAL TRIAL: NCT02169713
Title: A Phase 1 Study to Evaluate the Effect of Steady State Solifenacin and Mirabegron on the Steady State Pharmacokinetics of Tamsulosin HCl in Healthy Male Subjects
Brief Title: Study to Evaluate the Effect of Solifenacin and Mirabegron on the Tamsulosin Hydrochloride (HCl) Concentrations in Blood in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 178-CL-109; 2013-004230-15 (EudraCT Number)
Record Dates: First submitted 2014-06-05; First posted 2014-06-23 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Subjects; Pharmacokinetics; Drug-Drug Interaction (DDI)
Keywords: Healthy subjects; Mirabegron; Solifenacin; Tamsulosin HCl
MeSH Terms: interventions — mirabegron; Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Tamsulosin HCl alone (with matching placebo for solifenacin and mirabegron) then followed by tamsulosin HCl with solifenacin and mirabegron
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate; Drug: Tamsulosin HCl; Drug: Placebo
- Treatment Sequence 2 (Experimental): Tamsulosin HCl with solifenacin and mirabegron then followed by tamsulosin HCl alone (with matching placebo for solifenacin and mirabegron)
  Interventions: Drug: Mirabegron; Drug: Solifenacin succinate; Drug: Tamsulosin HCl; Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — Oral
  Other Names: Myrbetriq; Betmiga; Betanis
Drug: Solifenacin succinate — Oral
  Other Names: solifenacin; Vesikur; Vesicare
Drug: Tamsulosin HCl — Oral
  Other Names: Flomax
Drug: Placebo — Oral

SUMMARY:
The purpose of this study is to evaluate the effect of solifenacin and mirabegron on the concentrations of tamsulosin HCl after combined dosing. This study will also evaluate the safety and tolerability of the combined administration of solifenacin, mirabegron and tamsulosin HCl.

DETAILED DESCRIPTION:
This study is comprised of two study sequences with 2 investigational periods in each sequence. There will be a wash-out period between each investigational period. Patients will be admitted to the clinic until discharged after each investigational period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 to 30.0 kg/m2, inclusive. The subject weighs at least 50 kg [screening].
* Subject and their female spouse/partners who are of childbearing potential must be using a highly effective form of contraception consisting of 2 forms of birth control (one of which must be a barrier method) starting at screening and continue throughout the clinical study period and for 90 days after the final study drug administration.
* Subject must not donate sperm starting at screening and throughout the clinical study period and for 90 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participation in the present clinical study, defined as signing the informed consent form until completion of the last clinical study visit.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to solifenacin succinate, mirabegron, tamsulosin HCl or any components of the formulations used including sulfa allergies.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma-glutamyl transferase and/or total bilirubin [TBL]) above 1.5 of the upper limit of normal (ULN). In such a case the assessment may be repeated once [day-1].
* Subject has any clinically significant history of allergic conditions.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy, as judged by the Medical Investigator.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to day -2 (admission day).
* Subject has any clinically significant abnormality following the Investigator's review of the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or day -1.
* Subject has a mean pulse rate of < 50 or > 90 bpm; mean systolic BP < 90 mmHg or > 140 mmHg; mean diastolic BP < 60 mmHg or > 90 mmHg at day -1 (vital sign measurements taken in triplicate after subject has been resting in supine position for 10 min; pulse rate will be measured automatically).
* Subject has a mean QTc(F) interval of > 430 ms (> 450 for subjects aged 65 and above) at day -1. If the mean QTc(F) exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject has any clinical significant history of or risk of urinary retention, severe gastrointestinal condition (including toxic megacolon), myasthenia gravis or narrow-angle glaucoma, orthostatic hypotension.
* Subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease, or a family history of Long QT Syndrome.
* Subject uses any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies [e.g., St. John's Wort]) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day).
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit on day -2.
* Subject has a history of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit on day -2.
* Subject has consumed grapefruit (more than 3 x 200 mL) or marmalade (more than 3 times), star fruit, Seville oranges or Seville orange juice-containing products in the week prior to admission to the clinical unit until end of study visit (ESV), as reported by the subject.
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit regularly.
* Subject has significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinical unit admission on day -2.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis B core antibodies, hepatitis A virus antibodies (Immunoglobulin M), hepatitis C virus antibodies or human immunodeficiency virus 1 + 2 antibodies.
* Subject participated in any clinical study or has been treated with any investigational drugs within 28 days prior to screening.
* Subject is a vulnerable subject (e.g., subject kept in detention).
* Subject is an employee of the Astellas Group or Contract Research Organization involved in the clinical study.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter for tamsulosin HCl (plasma) in the absence and presence of solifenacin and mirabegron: Cmax | Day 14 in each investigational period
  Maximum concentration (Cmax)
Pharmacokinetic parameter for tamsulosin HCl (plasma) in the absence and presence of solifenacin and mirabegron: AUCtau | Day 14 in each investigational period
  Area under the curve over a dosing interval (AUCtau)

SECONDARY OUTCOMES:
Pharmacokinetic parameter for tamsulosin HCl (plasma): Ctrough | Days 11, 12 and 13 in each investigational period
  Concentration immediately prior to dosing at multiple dosing (Ctrough)
Pharmacokinetic parameter for tamsulosin HCl (plasma): tmax, CL/F, PTR | Day 14 in each investigational period
  Time after dosing when Cmax occurs (tmax), apparent total systemic clearance after single or multiple extra-vascular dosing (CL/F), Peak-through ratio (PTR)
Pharmacokinetic parameter for solifenacin and mirabegron (plasma): Ctrough | Days 11, 12 and 13 in each investigational period
  Concentration immediately prior to dosing at multiple dosing (Ctrough)
Pharmacokinetic parameter for solifenacin and mirabegron (plasma): Cmax, AUCtau, tmax, CL/F | Day 14 in each investigational period
  Maximum concentration (Cmax), Area under the curve over a dosing interval (AUCtau), Time after dosing when Cmax occurs (tmax), apparent total systemic clearance after single or multiple extra-vascular dosing (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Physician, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel International GmbH, Berlin, Germany